CLINICAL TRIAL: NCT03002714
Title: BLOOD PRESSURE REACTIVITY TO MENTAL STRESS IS ATTENUATED FOLLOWING RESISTANCE EXERCISE IN ELDERLY HYPERTENSIVE WOMEN
Brief Title: Blood Pressure Reactivity After Resistance Exercise in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ricardo Moreno Lima, Dr. (PhD), University of Brasilia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 307630/2013-7; 487622/2012-0 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2016-12-21; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Resistance Exercise Pressor and Neural Responses in Older Women
Keywords: Resistance Training; Psychological Stress; Aging; Hypertension; Autonomic Nervous System
MeSH Terms: conditions — Stress, Psychological; Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Performance of two resistance exercise sessions
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
The purpose of this study is to determine and compare the effects of two sessions of resistance exercise in blood pressure reactivity to a mental stress test in older hypertensive women.

ELIGIBILITY:
Inclusion Criteria:older hypertensive women -

Exclusion Criteria:subjects taking hormonal therapy; those with a history of metabolic, neurologic, or cardiovascular diseases other than HTN, those with a history of cardiovascular events; subjects with physical limitations; those with non-treated HTN; obesity (BMI ≥ 30.0); and subjects taking adrenergic inhibitors or non-dihydropyridinic calcium channel blockers.

-

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure reactivity to mental stress | 6 months

IPD SHARING:
Plan to Share IPD: No